CLINICAL TRIAL: NCT04659590
Title: An Exploratory Study Investigating the Potential of a Rectal Mucus Sample for Development of Biomarker Assays in Subjects With Gastrointestinal Diseases
Brief Title: Exploratory Study of Rectal Mucus for Diagnosing Disease
Acronym: ORI-EGI-02
Status: Completed | Type: Observational
Sponsor: Origin Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 263745
Record Dates: First submitted 2020-10-12; First posted 2020-12-09 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2022-08

CONDITIONS: Bowel Cancer; Bowel Disease; Genomic; Epigenetic Disorder
MeSH Terms: conditions — Intestinal Neoplasms; Intestinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Banked DNA retrieved from specimen taken from bowel lumen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The identification of patients with colorectal cancer is challenging as they present with a variable symptom profile and require invasive tests (colonoscopy) for diagnosis (through histological analysis of biopsies) and complimented by cross-sectional radiology, prior to commencement of treatment. The biopsy forms the basis of the diagnosis and management planning for a patient with colorectal cancer through the multidisciplinary team.

The biggest challenge currently faced in the management of colorectal cancer is the accurate identification of patients who present with various symptoms none of which are specific for bowel cancer. Currently the NICE referral guidelines are used to determine the appropriateness of referral pathway, i.e. Fast-Track/Two-Week Wait referral. A recent review of over 10000 referrals revealed a colorectal cancer diagnosis in 4.1% of referrals. Previous literature reports rates as high as 8%, but in series of cases with only 72-89% adherence to the referral guidance leading to at best 40% of all colorectal cases being diagnosed through this route. The remainder of colorectal cancers being diagnosed through the bowel cancer screening programme (NBCSP), non-two-week wait referrals and other processes such as emergency admissions. Inherently the Two-Week Wait pathway refers a large volume of "symptomatic patients" and it has become a "cancer exclusion pathway." Once cancer has been excluded, patients are often discharged back to General Practice, yet the patients often still have symptoms. The current Covid-19 pandemic has had a significant impact on the already pressed Two-Week pathway impacting on the reduction of endoscopic and radiological appointments available leading to delays in treatment. Each test performed in the diagnostic pathway has a significant financial, personal, and institutional resource profile.

It is our aim to develop a novel diagnostic device based upon the identification of genetic mutations and genomic alterations from material trapped in the rectal mucous layer allowing focused endoscopic assessment, confirmation/exclusion of cancer diagnosis from cross-sectional imaging in those unfit for endoscopic examination and identification of high-risk lesions (dysplasia). This would allow a greater triage, and focus colonoscopic services onto therapeutic procedures, improving overall care.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the fourth most common cancer overall worldwide contributing to 9.7% of global cancer burden. It affects 746,000 men (10% of all cancer cases) and 614,000 women (9.2% of all cancer cases) with most cases (55%) occurring in developed countries. Furthermore, in the UK, 42,300 new colorectal cancer cases are diagnosed each year making it the fourth most common cancer overall, and third most common in males and females. In addition, the incidence of colorectal cancer increased between 1991 and 2016 and is attributed to lifestyle, environmental changes, and aging populations. Although bowel cancer incidence has fallen in the UK in the past decade by 4%, the lifestyle risk factors remain. Moreover, the burden of CRC is expected to increase with 2.2 million new cases and 1.1 million deaths expected globally by 2030. In addition, significant challenges remain in managing disease burden.

In England, five-year overall survival for CRC is 58.4% which is lower than the US reported 60-65%. Further challenges remain due to the ageing demographic and advanced presentation of disease. Older patients, above age 75 years, make up 44% of new colorectal cancer diagnoses and an estimated 20-25% of CRC is diagnosed at the metastatic stage with an additional 25% of patients developing metastasis during their illness. As a result, CRC accounts for 8.5% of cancer related deaths worldwide with 16,300 deaths per year in the UK making it the second most frequent cause of cancer related deaths at 10%. Although survival is stage dependent with 92% survival for stage I, compared to 10% in stage IV, there has been an improvement in survival for the 60-69-year age group attributed to screening. Thus, CRC remains a prevalent challenge in cancer management emphasizing the need for early diagnosis.

Declining mortality due to improvements has been shown with early detection through screening and effective treatment. The UK CRC screening program relying on faecal detected occult blood (FOBT) and colonoscopy has led to 16% decline in overall mortality rate without affecting incidence. However, FOBT has reduced sensitivity for advanced adenomas and CRC which may improve with newly implemented immunochemical testing (qFiT). With the pressures on service from the Covid-19 pandemic, qFIT has been implemented into the Two-Week Pathway to attempt to stratify patients at highest risk of colorectal cancer and the NICE-qFiT Study publication is awaited.

Biomarkers are molecular patterns that can be used as a tool for early cancer detection and individualized CRC treatment. They can be divided into diagnostic, prognostic, or predictive categories. Thus, biomarkers provide utility at different stages of the disease to determine disease progression, recurrence, as well as providing a personalized indicator for therapeutic effectiveness.

Firstly, early diagnosis in asymptomatic patients remains a key target to achieve favourable survival outcomes through identification of early CRC as well as pre-malignant lesions including high risk polyps. This forms the basis of the National Bowel Screening Programme. The sensitivity for detecting CRC using current qFIT testing (100ng/mL) is 73.8% versus 92.3% for a stool-based DNA assay screening KRAS, aberrant NDRG4 and BMP3 methylation. Furthermore, qFIT testing sensitivity for advanced precancerous lesions is 23.8% versus 42.4% with stool DNA testing. Moreover, the rate of detection of polyps with high-grade dysplasia is 46.2% with qFIT testing verses 69.2% with stool DNA testing, whereas the detection rate of serrated sessile polyps measuring >1 cm is only 5.1% (qFIT) versus 42.4% with stool DNA sampling. These findings highlight the limits of current diagnostic screening and difficulty in establishing appropriate surrogate markers for early disease detection in asymptomatic individuals.

Current non-invasive screening stools are not sensitive to detect pre-cancerous lesions and regularly miss significant early CRC.

As outlined, the investigator currently have a low threshold in symptomatic patients for colonoscopy in these patients and further tools are required to support identifying early pre-malignant lesions (adenomas) and CRC .

The investigator knows from the recognition of the adenoma - carcinoma sequence and the impact of hyper- and hypomethylation that the local environment that there are a number of steps both in carcinogenesis and the associated risks.

At an epigenetic level, DNA methylation changes is one of the hallmark events in carcinogenesis, characterized by global hypomethylation and paradoxical gene-specific hypermethylation. Hypomethylation is primarily involved in chromosomal instability and global loss of imprinting, while gene-specific hypermethylation anchors to promoters, it causes transcriptional silencing of tumour suppressor genes and consequently sets the stage for neoplastic transformation. Deregulated DNA methylation is well known to be associated with CRC. The first evidence of DNA methylation contributing to CRC was presented, in which a global loss in DNA methylation was identified. Then, extensive efforts have been made in identifying aberrant hypermethylation in promoters of CRC-related suppressor genes, such as APC, SFRP2, SEPT, and CDH1. Remarkably, a near universal phenomenon that gene-specific hypermethylation occurred in both pre-neoplastic and neoplastic phase of colorectal cancer was observed. This might shed light on the process of tumorigenesis. However, few studies have defined precisely the hierarchy of methylation events during the transformation from normal epithelial cells to malignant cells in colorectal carcinogenesis.

It is becoming increasingly apparent that the occurrence of molecular alterations could be found not only in tumour tissue but also in histological normal-appearing tissue adjacent to the tumour. The presence of such molecular alterations in histological normal-appearing tissue is commonly known as field cancerization or field effect. This has been thought to constitute the earliest clone in the carcinogenesis process. In colorectal carcinogenesis, a few numbers of gene-specific hypermethylation events have been reported in normal-appearing colonic mucosa from CRC patients (such as APC, DKKI, MGMT, CDKN2A, and SFRP4). In addition, previous studies have also demonstrated the effect of aberrant DNA methylation on suppressor genes such as MINT1, MINT31, SLC5A8, and MGMT, during adenoma-carcinoma sequence. These findings suggest that the presence of field effect in methylation might be a useful intermediate biomarker in etiologic studies. A better understanding of when these epigenetic tags occur and how they take part in colorectal progression may represent a practical opportunity for colorectal cancer risk assessment. The use of a unique biological material capture device with genomic and epigenetic assessment of the retrieved specimen is the basis of the trial.

ELIGIBILITY:
Inclusion Criteria:

General inclusion criteria:

* aged 18 years or over
* be able to give voluntary, written informed consent to participate in the study

Exclusion Criteria:

* Subjects with confirmed collagenous colitis or symptoms that would make proctoscopic examination inappropriate, including acute anal fissure, symptomatic thrombosed haemorrhoids or obstructing anorectal tumours as determined by rectal examination
* Subjects with a previous history of cancer or who have previously received radiotherapy, chemotherapy or immunotherapy

The following populations will be included:

* Subjects with confirmed colorectal cancer
* Subjects with suspected colorectal cancer
* Subjects with known or suspected inflammatory bowel disease
* Known controls

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with known or suspected gastrointestinal disease(s).
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2019-11-06 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Stability of buffer transfer medium | through study, an average of 1 year
  Sample loss rate

SECONDARY OUTCOMES:
Comparison to qFiT test | through study, an average of 1 year
  Comparison to pathology identified
Comparison between tumour surface imprint and rectal mucous imprint | through study, an average of 1 year
  Comparison between tumour imprint surface and rectal mucous imprint

CONTACTS AND LOCATIONS:
Overall Officials: Jon Lacy-Colson, FRCS, Principal Investigator — Royal Shrewsbury Hospital
Locations (4):
- United Kingdom (4):
  - Royal Cornwall Hospital, Truro, Cornwall
  - John Radcliffe Hospital, Oxford, Oxfordshire
  - Royal Shrewsbury & Telford Hospitals NHS Trust, Shrewsbury, Shropshire
  - Royal Devon & Exeter NHS Foundation Trust, Exeter